CLINICAL TRIAL: NCT03703687
Title: Impact of a Gratitude-based Intervention on Patients and Caregivers in a Palliative Care Context: a Pilot Study
Brief Title: Impact of a Gratitude-based Intervention in Palliative Care (IPBG)
Acronym: IPBG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Mathieu BERNARD, Head of the Research Unit of the palliative and supportive care service, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPBG2018-2020
Record Dates: First submitted 2018-09-28; First posted 2018-10-12 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Palliative Care
Keywords: palliative care; gratitude; positive psychology

STUDY DESIGN:
Intervention Model Description: This clinical trial has a single arm: all the dyads will go through all the steps (apart from the qualitative assessment which are facultatives).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gratitude intervention (Experimental): The intervention will be proposed to both the patient and the caregiver and consists of two steps: the "gratitude letter" and the "gratitude visit". In the "gratitude letter", the individual writes about his feelings of gratitude through a letter, based on a written instruction. The "gratitude visit" consists of an extension of the gratitude letter where the writer of the letter (i) either personally reads the letter to the beneficent or (ii) gives it to him and asks him to read it in his presence or later in his absence.
  Interventions: Behavioral: Gratitude intervention

INTERVENTIONS:
Behavioral: Gratitude intervention — The intervention will be proposed to both the patient and the caregiver and consists of two steps: the "gratitude letter" and the "gratitude visit". In the "gratitude letter", the individual writes about his feelings of gratitude through a letter, based on a written instruction. The "gratitude visit" consists of an extension of the gratitude letter where the writer of the letter (i) either personally reads the letter to the beneficent or (ii) gives it to him and asks him to read it in his presence or later in his absence.
  Other Names: gratitude letter; gratitude visit

SUMMARY:
This is a pilot study consisting of mixed-methods, pre-post evaluation of a gratitude intervention (gratitude letter and visit) on palliative care patients and their caregivers.

DETAILED DESCRIPTION:
Study background and aims:

Gratitude, defined as an "other-oriented" emotion, has shown to impact significantly on many relevant dimensions for palliative care (e.g. well-being, psychological distress and the quality of relationships). Various psychological interventions focused on the enhancement of the feeling of gratitude have been developed and assessed but mostly in non-clinical populations and never taking into account the relationship dimension as an outcome.

The fact that the relational component has never been addressed in interventional studies is all the more surprising since several experimental and non-clinical studies have clearly shown an association between gratitude and feeling of social affiliation, relational commitment, satisfaction with relationships or partner reciprocal maintenance behaviours. These results appear to be very promising for palliative care since interpersonal (and particularly familial) relationships are crucial for palliative care patients: the relational sphere represents a major predictor contributing to both their meaning in life and their quality of life. We hypothesize that considering this concept in palliative care could benefit both the patients and their relatives.

Thus, the purpose of this research is to conduct a pilot study before a possible randomized controlled multicenter trial whose final aim will be to examine whether a gratitude-based intervention in a palliative care setting can increase the quality of life and the quality of the relationship of patients and their caregivers and decrease their psychological distress and burden.

The specific aims of this pilot study are:

(i) to realize a cross-cultural translation of outcome measures that are not yet available in French (ii) to establish the feasibility of the study design (iii) to investigate the appropriateness of the gratitude concept and the gratitude-based intervention in the palliative care context, and finally (iv) to explore the sensitivity to change of our selected measures in order to calculate a sample size.

Procedure and measures:

Quantitative data will be collected at baseline (T0) and post-intervention (T1) with validated questionnaires. The intervention will last for one week. Five to ten days after T1, qualitative data will be collected from semi-structured interviews with the participants and from the content of the gratitude letters to explore their representations of the gratitude concept and their perception of the intervention.

The intervention includes the following steps:

1. Patients and caregivers recruitment: The clinical team (treating physician or advanced practice nurse) at each recruitment site will identify 10 patient-caregivers dyads. A research collaborator will then be in charge of giving information and get consent
2. Data collection at T0: Before the intervention, patients and their caregivers who agreed to participate will meet the research collaborator to fill quantitative questionnaires.
3. Intervention - 1-week duration: The intervention will be proposed to both the patient and the caregiver and consists of two steps: the "gratitude letter" and the "gratitude visit". In the "gratitude letter", the participant (at least one of the patient or the caregiver) writes about his feelings of gratitude through a letter, based on a written instruction. The "gratitude visit" consists of an extension of the gratitude letter where the writer of the letter (i) either personally reads the letter to the beneficent or (ii) gives it to him and asks him to read it in his presence or later in his absence.
4. Data collection at T1: 5 to 10 days after the intervention itself, the patient and the caregiver, will meet with the research collaborator again to participate to a second quantitative assessment, similar to T0.
5. Qualitative assessment: 5 to 15 days after T1: This part is facultative. During the qualitative interviews, the following topics will be explored: their meanings of the term "gratitude"; experiences of gratitude; their experience of the intervention itself; obstacles and facilitators of the intervention; the impact of the intervention for themselves and for their relationship.

ELIGIBILITY:
Only patients fulfilling all of the following inclusion criteria are eligible for the study:

* Age >18
* progressive disease
* reduced life expectancy
* enrolment in palliative care
* stable state for the previous 24h assessed by the physician or the nurse in charge of the patient
* informed consent signed by patient
* For each patient, the identification of a close family or friend caregiver (fulfilling the below criteria*) and who accepts to participate in the trial (by signing an informed consent)

In this research, a caregiver is defined as "a person who devotes time to help a family member or a friend affected in her/his health or autonomy. The caregiver assures, in a non-professional and regular way, a presence and a support to help her/him in his difficulties and assures her/his safety. The caregiver can be a friend, a family member or a neighbour" (Vaud canton definition). This definition will be the basis for the palliative patient to identify his caregiver.

The presence of any one of the following exclusion criteria will lead to exclusion of the patient:

* Person completely isolated socially, no family or friend caregiver identified
* Significant cognitive or psychiatric disorders which would affect the ability to give informed consent for this research
* Severe communication problems (foreign language, deafness, etc.).

Only caregivers fulfilling all of the following inclusion criteria are eligible for the study:

* Age >18
* Identified as the caregiver by the palliative patient (see above)
* prior agreement of the patient for the participation of the caregiver

The presence of any one of the following exclusion criteria will lead to exclusion of the caregivers:

* Psychiatric and cognitive disorders which would affect the ability to give informed consent for this research based on the information reported by the clinical team in charge of the patient and the personal evaluation of the research collaborator.
* Communication problems (foreign language, deafness, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Change in relationship quality for patients and caregivers | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  The quality of the relationship between the palliative patient and his/her caregiver will be measured with the Couple Satisfaction Index (CSI-4; "total score" range from 0 to 21, higher scores indicating a better quality of relationship).
Change in relationship quality for patients and caregivers | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  The quality of the relationship between the palliative patient and his/her caregiver will be also measured with the Positive Negative Relationship Quality Scale (PNRQ; "positive subscale" range from 0 to 48 and "negative subscale" range from 0 to 48, with higher scores indicating higher quality of relationship).

SECONDARY OUTCOMES:
Change in subjective quality of life for patients | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  The quality of life will be measured with the McGill Quality of Life scale Revised version (MQOL-R; all subscales range from 0 to 10: "global quality of life", "physical", "psychological", "existential", "relationships", and "total score", with higher scores indicating higher quality of life)
Change in subjective quality of life for caregivers | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  The quality of life will be measured with the Quality of Life in Life-Threatening Illness - Family Carer Version 2 (QOLLTI-F V2; all subscales range from 0 to 10: "global quality of life", "environment", "patient condition", "own condition", "outlook", "quality of care", "relationships", "financial worries", and "total score", with higher scores indicating higher quality of life)
Change in psychological distress for patients | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  Psychological distress will be measured with the Hospital Anxiety and Depression Scale (HADS; "total score" range from 0 to 42; "anxiety subscale" from 0 to 21, and "depression subscale" from 0 to 21, with higher scores indicating higher distress)
Change in psychological distress for caregivers | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  Psychological distress will be measured with the Brief Symptom Inventory 18 (BSI 18; "total score" range from 0 to 72, "somatic subscale" range from 0 to 24, "depression subscale" range from 0 to 24, "anxiety subscale" from 0 to 12; and "panic subscale" from 0 to 12, with higher scores indicating higher distress).
Change in burden for patients | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  Burden will be measured with the Self Perceived Burden Scale (SPBS, "total score" range from 10 to 50, with higher scores indicating higher burden).
Change in burden for caregivers | Baseline approx. 5 days before intervention; post-intervention approx.10 days after intervention
  Burden will be measured with the 10-item short version of the Burden Scale for Family Caregivers (BSFC-s, "total score" from 0 to 30, with higher score indicating higher burden).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Bernard, Principal Investigator — Palliative and Supportive care service of the Centre Hospitalier Universitaire Vaudois
Locations (3):
- Switzerland (3):
  - Rive-Neuve Foundation, Blonay, Canton of Vaud
  - Lausanne University hospital, Palliative and supportive care service, Lausanne, Canton of Vaud
  - Fribourg University hospital, Unité et Accueil de jour de soins palliatifs, Fribourg

IPD SHARING:
Plan to Share IPD: Undecided
Undecided up to now